CLINICAL TRIAL: NCT01715766
Title: VIPER: Veterans Integrated Pain Evaluation Research- Molecular Subtypes of Chronic Pain Syndromes
Brief Title: VIPER: Veterans Integrated Pain Evaluation Research
Acronym: VIPER
Status: Completed | Type: Observational
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: 360806-15
Record Dates: First submitted 2012-10-17; First posted 2012-10-29 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Pain
Keywords: Proteomics study; biomarker study of pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood draw will consist of, two BD™ P100 tubes (2x8.5mL=17mL) where the plasma will be separated by centrifuge then placed in a -80ºC freezer. Two RNA tubes (2 x 2.5mL=5mL) and one DNA tube (8.5mL) will be place first, in a -20ºC freezer for 24-36 hours then moved to a -80ºC freezer. All the blood samples will remain in a -80ºC freezer at the Department of Clinical Investigation(DCI) laboratory until they are sent to Duke University after every 8 subjects.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to learn about the causes of different types of pain that can occur in people who have had an amputation. By gathering information through blood tests, photographs, a nerve test, and questionnaires, we hope to de-code how each individual's special characteristics affect the type and amount of pain they experience in their amputated limb.

DETAILED DESCRIPTION:
Studies have already shown that pain following amputation might be caused by differences in a person's genes. This study may help us find out how genes affect the way you feel pain and why you may feel more or less or different kinds of pain than another person with a similar amputation. What we learn in this research study may lead to discoveries as to why some painkillers work better for some people than others.

ELIGIBILITY:
Inclusion Criteria:

* Male and female active duty military personnel age 18 years and older undergoing treatment at WRAMC and future WRNMMC with the diagnosis of post injury amputation of 1 limb, more than 3 but less than 18 months prior to enrollment. In particular, phantom limb pain patients will be included

Exclusion Criteria:

* Severe Traumatic Brain Injury (Primary major head trauma and diagnosis of traumatic brain injury resulting in documented, permanent or prolonged cognitive deficits that would preclude participation in the study (i.e. decreased intellectual capacity, marked memory deficits, or inability to communicate verbally or in writing)
* Significant cognitive deficits that would preclude participation in the study.
* Substantial hearing loss without alternative means of communication.
* Documented spinal cord injury with permanent or persistent deficits.
* Diagnosis of fibromyalgia or other chronic pain syndrome such as chronic headaches.
* Evidence of ongoing tissue damage pain, infection, bone spur, or poorly fitting prosthesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female active duty military personnel age 18 years and older presenting with the diagnosis of amputation of 1 limb in the previous 18 months. At least 3 months must have passed since the first amputation procedure.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Proteomics | 1 day
  To determine which proteins represent circulating qualitative and quantitative biomarkers of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States